CLINICAL TRIAL: NCT05921734
Title: A Randomized Controlled Study of Ablation Pursuing Atrial Fibrillation Termination as a Procedural Endpoint Versus Prespecified Ablation Strategy Followed by Cardioversion in Patients With Persistent Atrial Fibrillation
Brief Title: A Randomized Controlled Study of Ablation Pursuing Atrial Fibrillation Termination as a Procedural Endpoint in Patients With Persistent Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Xu Liu, Principal Investigator, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAPT-AF
Record Dates: First submitted 2023-06-10; First posted 2023-06-27 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2023-06

CONDITIONS: Atrial Fibrillation; Cathter Ablation; Endpoint
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AF-termination Group (Experimental)
  Interventions: Procedure: AF-termination Group
- Prespecified-ablation Group (Active Comparator)
  Interventions: Procedure: Prespecified-ablation Group

INTERVENTIONS:
Procedure: AF-termination Group — Each center completes the ablation according to the above ablation procedure. The choice of ablation strategy is not restricted, but efforts should be made to achieve termination of AF during the ablation procedure. If cannot terminate AF for safety or other reasons involving difficulties to remap AFEGM or creating a complete conduction block despite the operator's best efforts, then direct current conversion (DCCV) was performed.
  Arms: AF-termination Group
Procedure: Prespecified-ablation Group — Each center completes the prespecified ablation according to the above ablation procedure. Although there is no restriction on the choice of ablation strategy, Ablation must be performed following the PVI plus strategy, which can be combined with one or more additional ablation procedures, but each ablation must achieve its own endpoints, such as bidirectional block of linear damage, posterior wall isolation, etc. After completing the preset ablation steps, DCCV will be performed. If AF is terminated after or during ablation, it is also considered the endpoint of ablation in this group, but the preset ablation steps must be completed.
  Arms: Prespecified-ablation Group

SUMMARY:
This is a prospective, randomized, multi-center trial that aims to investigate whether termination of atrial fibrillation can be used as an ablation endpoint for persistent atrial fibrillation (PersAF). Eligible patients who provided consent were randomly assigned to one of two groups: the AF-termination group (whose ablation endpoint was the pursuit of AF-termination) or the prespecified-ablation group (whose ablation endpoint was prespecified ablation followed by electrical cardioversion).

ELIGIBILITY:
Inclusion Criteria:

1. . Age 18-80 years old.
2. . Patients undergoing a first-time ablation procedure for PersAF.
3. . Diagnosed as persistent AF according to the latest clinical guidelines.
4. . Ineffective or intolerable to ≥1 anti-arrhythmia drug treatment.
5. . Patients must be able and willing to provide written informed consent to participate in this study.

Exclusion Criteria:

1. . Uncontrolled congestive heart failure;
2. . History of severe valve disease and/or prosthetic valve replacement;
3. . Myocardial infarction or stroke within 6 months;
4. . Severe congenital heart disease;
5. . EF <35%;
6. . Contrast agent allergy;
7. . The use of anticoagulant drugs is contraindicated;
8. . Severe lung disease;
9. . Left atrial thrombus confirmed by preoperative esophageal ultrasound;
10. . Contraindications for cardiac catheterization;
11. . Prior left atrial ablation (surgical or catheter);
12. . Have performed any cardiac surgery within 2 months;
13. . Poor general health;
14. . Life expectancy < 12 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
freedom from any documented atrial arrhythmia - atrial fibrillation (AF), atrial tachycardia (AT), or atrial flutter (AFL) - of more than 30 seconds, excluding the initial 3 months blanking period | Time Frame: 12 months
  All patients included in the study had no incidence of Atrial fibrillation (AF), atrial tachycardia (AT) or Atrial flutter (AFL) at 12 months after ablation, excluding the initial 3-month blank period

SECONDARY OUTCOMES:
freedom from AF/AT after a single procedure without AADs (excludes the blanking period) | Time Frame: 12 months
  All patients included in the study had no incidence of AF/AT after a single procedure without AADs at 12 months after ablation excluding the initial 3-month blank period
freedom from AF/AT after a single procedure with or without anti-arrhythmic medications (excludes the blanking period) | Time Frame: 12 months
  All patients included in the study had no incidence of freedom from AF/AT after a single procedure with or without anti-arrhythmic medications at 12 months after ablation excluding the initial 3-month blank period
any documented AF episode lasting more than 30 seconds after the blanking period without anti-arrhythmic drugs (AADs) treatment | Time Frame: 12 months
  All patients included in the study had no incidence of any documented AF episode lasting more than 30 seconds after the blanking period without anti-arrhythmic drugs (AADs) treatment at 12 months after ablation, excluding the initial 3-month blank period
freedom from any AT episodes lasting more than 30 seconds after the blanking period without AADs after a single procedure | Time Frame: 12 months
  All patients included in the study had no incidence of any AT episodes lasting more than 30 seconds after the blanking period without anti-arrhythmic drugs (AADs) treatment at 12 months after ablation, excluding the initial 3-month blank period
procedural details | Time Frame: 12 months
  All patients' procedural details: including procedure time, mapping time, fluoroscopy time, ablation time.
incidence of periprocedural adverse events | Time Frame: 12 months
  All patients' periprocedural adverse events including：ascular- significant groin，haematoma, pseudoaneurysm, AV fistula，Cardiac perforation，Pericardial effusion/ tamponade，Pericarditis，Pneumothorax/ haemothorax，Phrenic nerve injury，Periprocedural cerebrovascular accident - including air embolism，Esophageal injury - perforation / atrio-esophageal fistula，Pulmonary vein stenosis，Major bleeding event -including retroperitoneal bleeding，Heart block，Death

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Mu Qin, Shanghai
  - Shanghai Chest Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided